CLINICAL TRIAL: NCT07001085
Title: A Prospective Randomized Trial Assessing the Impact of ctDNA Testing in Patients After Liver Resection or Transplantation Due to Metastases From Colorectal Cancer or Hepatocellular Carcinoma (HCC) on Treatment Strategies and Long-term Survival"
Brief Title: ctDNA Monitoring in Patients With HCC and mCRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Oskar Kornasiewicz, Associate Professor, MD, PhD Oskar Kornasiewicz, Medical University of Warsaw
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1WB1; 2023/ABM/01/00068 (Other Grant/Funding Number: Medical Research Agency)
Record Dates: First submitted 2025-05-09; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-01

CONDITIONS: HCC - Hepatocellular Carcinoma; Colorectal Cancer Metastatic
Keywords: ctDNA; MRD; CRC; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study Group - Colorectal Cancer with Liver Metastases (Other): Patients with metastatic colorectal cancer to the liver. Tumor tissue obtained during surgery is subjected to DNA extraction and Next-Generation Sequencing (NGS) to identify oncogenic mutations. Blood samples are collected one day before surgery, one month, and six months after surgery. Plasma is separated from blood to isolate circulating tumor DNA (ctDNA), which is then tested using droplet digital PCR (ddPCR) to detect the mutations previously identified by NGS.
  Interventions: Diagnostic Test: Tumor Tissue Collection and NGS; Other: Blood Collection for Plasma ctDNA; Diagnostic Test: ctDNA Mutation Analysis via ddPCR
- Study Group - Hepatocellular Carcinoma (Other): Patients with hepatocellular carcinoma. Tumor tissue collected during surgery is analyzed using NGS to identify oncogenic mutations. Blood samples are collected at the same three time points. Plasma-derived ctDNA is tested using ddPCR for the previously detected mutations.
  Interventions: Diagnostic Test: Tumor Tissue Collection and NGS; Other: Blood Collection for Plasma ctDNA; Diagnostic Test: ctDNA Mutation Analysis via ddPCR
- Control Group - Colorectal Cancer with Liver Metastases (Other): Patients with metastatic colorectal cancer to the liver meeting control group criteria. Blood samples are collected one day before surgery, one month, and six months after surgery. Plasma is separated and stored, but no NGS or ddPCR analyses are performed.
  Interventions: Other: Blood Collection for Plasma ctDNA
- Control Group - Hepatocellular Carcinoma (Other): Patients with hepatocellular carcinoma meeting control group criteria. Blood is collected at three predefined time points. Plasma is separated and stored. No molecular or genetic testing is conducted on these samples.
  Interventions: Other: Blood Collection for Plasma ctDNA

INTERVENTIONS:
Diagnostic Test: Tumor Tissue Collection and NGS — Tumor tissue is collected during surgery and used for DNA extraction. Next-Generation Sequencing (NGS) is performed to identify oncogenic mutations.
  Arms: Study Group - Colorectal Cancer with Liver Metastases; Study Group - Hepatocellular Carcinoma
Other: Blood Collection for Plasma ctDNA — Blood is collected at three time points: one day before surgery, one month, and six months after surgery. Plasma is separated and used for further molecular analysis or storage.
Diagnostic Test: ctDNA Mutation Analysis via ddPCR — Circulating tumor DNA (ctDNA) is isolated from plasma samples. Mutations previously identified by NGS are quantitatively analyzed using droplet digital PCR (ddPCR).
  Arms: Study Group - Colorectal Cancer with Liver Metastases; Study Group - Hepatocellular Carcinoma

SUMMARY:
"Liquid biopsy" is a collective term that refers to the analysis of cancer-derived biomarkers isolated from the biological fluids of cancer patients. The analysis of these blood components can be used for early cancer detection, staging, prognosis, drug resistance monitoring, and minimal residual disease (MRD) monitoring. The "liquid biopsy" is based on the fact that cancer cells release their DNA into the bloodstream, known as ctDNA (circulating tumor DNA). A sample of the patient's peripheral blood is sufficient to test ctDNA. There have been many studies in the literature on the usefulness of liquid biopsy in the treatment of various malignancies, such as breast cancer, prostate cancer, and colorectal cancer. However, this has been a lack of prospectively obtained data analyzing the impact on the ctDNA assessment of the progression and recurrence of the primary disease or the type of treatment applied to improve long-term survival. The ctDNA test is not a widely recognized technology for assessing the progression of neoplastic disease.

Aim of the study/research hypothesis: the aim of the project is to clinically validate the value of the ctDNA test as a tool for early diagnosis of recurrence, assessment of cancer progression, the prognosis of treatment effects, and monitoring of therapy in patients with primary liver HCC or colorectal cancer metastases.

Description of the methodology: The main objective of the work will be achieved through the implementation of specific objectives: 1) Recruitment of 300 patients, including 100 patients with colorectal liver limited metastasis, 100 patients with hepatocellular carcinoma (HCC) and 100 patients in the control group who will be qualified for liver resection or transplantation, and in whom ctDNA level testing will not be tested. 2) Taking blood samples from the patients. The detection of ctDNA requires only the collection of 10 ml of the patient's blood and the collection of specimens from the tumor after resection. Blood will be collected before, one month, and 6 months after surgery during routine oncology check-ups. Tumor specimens will be taken from the backside table and sent for final histopathological examination. Control "follow-up" will take place for 18 months from the first ctDNA blood collection.

Based on the collected material, genetic analysis will be performed. In the first stage, a tumor section taken during liver resection, and DNA from the patient's blood will be analyzed the molecular (genetic) signature of the patient's tumor will be determined and several genetic changes characteristic of the change will be selected. Thereafter, the presence of the selected genetic variants will be assessed qualitatively and quantitatively in the pre-operative blood sample and all subsequent post-operative blood samples.

The investigators assume that in a blood sample taken 4 weeks after surgery, ctDNA should be undetectable or detected at a low level. In order to assess the change in the level of ctDNA in the postoperative period, a third examination will be performed - 6 months after the operation. Any level of detected ctDNA will be considered significant.

Each increase in the level of the analyzed mutations will indicate the potential progression of the disease. The results of molecular analyzes will be correlated with the assessment of imaging tests and the level of tumor markers performed as part of routine oncological control.

This is a prospective observational study with a defined study group. These are patients with colorectal cancer metastases limited to the liver, i.e. stage IV of the cancer process, or patients with hepatocellular carcinoma (HCC) qualified for radical surgery or liver transplantation. Patients in the control group (without ctDNA tests) will be treated in accordance with the best clinical knowledge and accepted international recommendations.

The statistical analysis of the results will use the SAS (Statistical Analysis System) software, considering the Kaplan-Meier method, log-rank tests, Cox proportional hazards regression, and logistic regression.

The investigators hypothesize that the use of ctDNA will enable the identification of early disease progression or will identify patients with the highest risk of recurrence. In addition, it will improve the supervision of diseases and enable possible modification of treatment in patients with stage IV colorectal cancer or patients after liver resection or transplantation for HCC. In the future, oncological prevention will consist in blood tests, which will enable early detection of even those cancers that show symptoms only at an advanced stage, which will potentially improve the effectiveness of treatment.

DETAILED DESCRIPTION:
Health problem Hepatocellular carcinoma (HCC) is the most common primary malignant tumor of the liver. It is estimated that it accounts for 80-90% all cases of liver cancer. Liver cancer is one of the faster growing and worse prognosis cancers. It constitutes approximately 5.4% of all malignant tumors.

Colorectal cancer (CRC) is currently the third most common cancer in the world and in Poland. Every year in the Polish population about 20,000 people will be diagnosed with colorectal cancer. Most of them will be diagnosed in the advanced stage IV of the disease. About 50% of CRC patients will develop liver metastases during the natural course of disease progression. Surgery for liver metastases is the only potential treatment. Even after tumor resection surgery, the disease may continue to develop even if the patient is undergoing chemotherapy.

Furthermore, the accuracy and sensitivity of pathological and imaging methods for disease progression or molecular identification of residual disease (MRD) are limited, while when the specificity and clinical diagnostic utility of serum markers (CEA) is poor. CT/MRI/PET being part of the standard surveillance program increases ability to detect recurrences, but are not sensitive enough for small lesions, especially in patients after liver resection or modern chemotherapy, i.e. targeted therapy. Most patients have no measurable disease based on imaging until an obvious recurrence occurs. Often it is too late for any intervention. Each recurrence of the disease is also a failure of the chemotherapy. In addition, second line chemotherapy is less likely to work success in terms of long-term patient survival. Therefore, there is an urgent need to improve approaches to long-term non-invasive tumor monitoring and predict recurrence earlier than standard imaging, and to evaluate the effect of surgical intervention and chemotherapy, especially in stage IV cancer.

The awarding criterion - HCC is a rare disease. Awarding criterion - the area of surgery and diagnostics.

In the case of patients with colorectal cancer, the target group of patients to be included in the study are patients over 18 years of age with metastases of colorectal cancer. Colon limited to the liver, with no history of cancer other than colorectal cancer. The study will include synchronous and metachronous metastases according to: new definition.

In the case of hepatocellular carcinoma (HCC), the target group is patients with resectable HCC, in the case of liver resection or unresectable HCC in the case of liver transplantation. The study will include patients with or without cirrhosis. Qualification for liver transplantation and indication for transplantation liver disease will be taken into account, among others, using the French model of HCC (calculator), which takes into account the size and number of lesions and the AFP level.

Patients with or without cirrhosis will be qualified for liver resection. The group will include patients from the age of 18 to the age of 75 in the case resection and all patients qualified for liver transplantation at the liver transplantation qualification meeting.

Patients with completely removed primary tumor in the large intestine will be in the study group.

Chemotherapy is not an indication for the study. According to treatment standards, the vast majority of patients with colorectal cancer and/or metastases will undergo treatment chemotherapy. Currently, not enough scientific research has been conducted to determine how and whether chemotherapy administered to patients affects the results ctDNA. Additionally, the study assumes that patients will be covered by the standard of care in this group of patients.

Patients with extrahepatic lesions will not be included in the study. Patients with rapid disease progression on chemotherapy with a 6-month survival period uncertain will not be included in the research. Patients older than 75 years of age will also not be included in the study.

Patients undergoing steroid therapy and diagnosed with autoimmune diseases will not be included in the study.

The goal of surgical treatment is to achieve R0 resection of all liver metastases. Patients after liver resection with radiologically visible recurrence will undergo treatment further treatment according to the decision of the oncology team. Hepatic and extrahepatic recurrence does not exclude the patient from the study.

Detailed treatment protocol

1. Qualification of the patient for liver resection or transplantation. Assessment of patients at an oncology consultation.
2. Obtaining informed consent to participate in the study.
3. Randomization of patients in a 2:1 ratio by drawing a code indicating ctDNA testing (control group - without ctDNA testing)

3. Assessment of the patient immediately before surgery.

a. Physical and subjective examination. i. Assessment of quality of life using the Polish version of the EORTC QLQ-C30 form b. Performing laboratory and imaging tests in accordance with local protocol. i. Biochemical tests ii. Imaging tests 4. Collecting 10ml of blood for gDNA and ctDNA testing along with routine preoperative blood collection.

5. Surgery 6. Liver resection or orthotopic liver transplantation from a deceased donor. 8. Monitoring the patient in the surgical intensive care unit. 9. Monitoring the patient in the general room at the Department of General, Transplantation and Liver Surgery.

10. Discharge of the patient home and completion of surgical treatment. 11. Monitoring the patient in the general room of the Hepatology Clinic in the case of transplantation or in the Polyclinic in the case of liver resection.

12. Transplantation/surgical outpatient clinic: Assessment on the 30th day (with a deviation of 2-3 days) after surgery in terms of the occurrence of postoperative complications, assessment general examination of the patient and 2 taking a blood sample for ctDNA testing.

13. Transplant/surgical outpatient clinic: Assessment in the 6th month (with a deviation of a few days) after surgery in terms of the patient's general condition and possible recurrence cancer process, taking a third blood sample for ctDNA testing. 14. Transplant/surgical outpatient clinic: Monitoring the cancer process and assessing patients one year after resection/transplantation.

16. End of the observation period of patients 12 months after the last collection

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years of both sexes;
* patients with synchronous or metachronous metastases of colorectal cancer limited to the liver after complete removal of the primary lesion from the intestine qualified for liver resection or transplantation;
* or patients with resectable or unresectable HCC scheduled for liver resection or transplantation
* no history of other cancers;
* negative virological status in the case of mCRC;
* In the case of mCRC - patient after any type of liver surgery (staged, ALPPS, multi-site resection)
* Patient with or without neoadjuvant chemotherapy compatible with established adjuvant therapy

Exclusion Criteria:

* age under 18 and over 75;
* pregnancy
* patients with extrahepatic metastases visible in imaging studies;
* metabolic and autoimmune diseases or chronic immunosuppressive treatment other than in the group of patients after liver transplantation due to HCC;
* positive virological status, excluding the group of patients with HCC;
* history of other cancer;
* Chronic steroid therapy and diagnosed active autoimmune diseases
* Patient after radiotherapy
* Patient participating in other clinical trials of oncological and non-oncological drugs
* Patients legally incapacitated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the clinical value of ctDNA level | One day before surgery - first day of enrollment
  Assessment of the ctDNA concentration one day before surgery.
Assessment of the clinical value of ctDNA level | From enrollment to 30 days after a surgery.
  Assessment of the ctDNA concentration one month after surgery
Assessment of the clinical value of ctDNA level | From enrollment to 6 months after a surgery.
  Assessment of the ctDNA concentration 6 months after surgery.
Assessment of the mutational status of patient cancer | From enrollment to 6 months after a surgery.
  Determining the mutation status of the patient's cancer tissue by performing next-generation sequencing
Assessment of the mutational status of patient cancer | From enrollment to 6 months after a surgery.
  Determining the mutation status of the patient's cancer by performing ddPCR reaction.
Assessment of the mutational status of patient cancer 30 days after surgery | From enrollment to 6 months after a surgery.
  Determination of mutation status in plasma, 30 days after the patient's surgery by performing ddPCR reaction. This study aims to determine the rate of tumor recurrence.
Assessment of the mutational status of patient cancer 6 months after surgery | From enrollment to 6 months after a surgery.
  Determination of mutation status in plasma, 6 months after the patient's surgery by performing ddPCR reaction. This study aims to determine the rate of tumor recurrence.

SECONDARY OUTCOMES:
Assessment of quality of life | From enrollment to 4 years after a surgery.
  Assessment of quality of life using the Polish version of the EORTC QLQ-C30 form. The statistical analysis of the results will use the SAS (Statistical Analysis System) software, considering the Kaplan-Meier method, log-rank tests, Cox proportional hazards regression, and logistic regression.
Comparative evaluation of imaging results with molecular results | From enrollment to 4 years after a surgery.
  Evaluation of alpha-fetoprotein (AFP), carcinoembryonic antigen (CEA), and Ca19-9 antigen levels and their comparison with ctDNA results

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Stokłosa, Professor, Principal Investigator — tomasz.stoklosa@wum.edu.pl
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR